CLINICAL TRIAL: NCT02933541
Title: Central Arterial Pressure Changes With Use of Regional Anesthesia in Obstetric Patients
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Niraj R. Chavan, MD, MPH, MD, St. Louis University
Other Study IDs: 27440
Record Dates: First submitted 2016-09-12; First posted 2016-10-14 (Estimated); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Central Blood Pressures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Plan to monitor central arterial pressure in women who are undergoing spinal anesthesia for cesarean delivery or epidural anesthesia for vaginal delivery.

DETAILED DESCRIPTION:
Subjects will be screened as they are admitted to the maternity care floor (5th floor St. Mary's Hospital). Subjects will be approached if they are desiring regional anesthesia.

The subject will have an additional blood pressure cuff placed on the arm that anesthesia is not using for their blood pressure cuff. Central arterial pressure will be measured from the cuff:

* Prior to regional anesthesia placement
* Every 15 minutes for 1 hour
* Every 30 minutes for 2 hours Routine sphygmomanometer measurements will also completed at the above times. These are all study procedures.

Anesthesia will use their usual protocol for blood pressure monitoring and management during placement of, and after the procedure. No changes in patient management will be made based upon the central arterial pressure as the guidelines were developed with routine brachial pressure.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Planned regional anesthesia

Exclusion Criteria:

* Multiple pregnancy
* Emergent cesarean delivery
* Irregular heart rhythms or arrhythmias
* Peripheral arterial disease, leg artery disease
* Reynaud's phenomena
* Intense cold/hypothermia
* If there is a wound at location of where central arterial cuff would be placed or tonometer for carotid assessment
* Severe tachycardia (>120)
* Greater than 1st degree heart block
* Congestive heart failure or heart disease
* Inability to adequately monitor BP
* Use of magnesium sulfate

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women who are admitted to our obstetrics ward and are planning on receiving regional anesthesia will be approached.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Amount of change in central arterial pressure in obesity. | 3 hours
  To determine if women who are obese undergo a larger change in their central arterial pressure than is seen by routine brachial cuff assessment, and if this effect is dependent on the level of obesity.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No